CLINICAL TRIAL: NCT04281628
Title: Comparison Between Low-dose Ketamine Infusion and Intravenous Morphine Infusion for Analgesia in Laparotomy Myomectomy: A Double-blind, Randomized, Controlled Clinical Trial
Brief Title: Comparison Between Low-dose Ketamine Infusion and Intravenous Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: I-190414
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Ketamine
Keywords: Ketamine; Morphine; Laparotomy Myomectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): control group: where normal saline will be administered as a loading dose then infused with same rate of another group, throughout the whole surgery.
  Interventions: Drug: Control group
- ketamine group (Active Comparator): Ketamine group: will be administered ketamine in a loading dose of 0.2 mg/kg over 5 min pre incision followed-by an infusion at 0.2 mg/kg/h until the end of surgery.
  Interventions: Drug: Ketamine group:

INTERVENTIONS:
Drug: Ketamine group: — Ketamine group: will be administered ketamine in a loading dose of 0.2 mg/kg over 5 min pre incision followed-by an infusion at 0.2 mg/kg/h until the end of surgery.
  Arms: ketamine group
Drug: Control group — where normal saline was administered as a loading dose then infused with same rate of another group, throughout the whole surgery.
  Arms: Control group

SUMMARY:
Ketamine is an antagonist of N-methyl-d-aspartate (NMDA) receptor that not only abolishes peripheral afferent noxious stimulation, but it may also prevent central sensitization of nociceptors as shown in animal studies with excellent analgesic property even in subanesthetic doses. It is readily available and is being used currently, even by non-Anesthesiologists, to provide "sedation" for minor procedures.(.. Low-dose ketamine infusion in the perioperative period has shown to produce analgesia and decrease the requirements of opioid analgesics.. In obstetrics, it is being used as an adjunct to an inadequately functioning spinal anesthesia for caesarean section, as an induction agent for cesarean section and also to provide analgesia during labor in intermittent boluses.

DETAILED DESCRIPTION:
Ketamine is an antagonist of N-methyl-d-aspartate (NMDA) receptor that not only abolishes peripheral afferent noxious stimulation, but it may also prevent central sensitization of nociceptors as shown in animal studies with excellent analgesic property even in subanesthetic doses. It is readily available and is being used currently, even by non-Anesthesiologists, to provide "sedation" for minor procedures.(.. Low-dose ketamine infusion in the perioperative period has shown to produce analgesia and decrease the requirements of opioid analgesics.. In obstetrics, it is being used as an adjunct to an inadequately functioning spinal anesthesia for caesarean section, as an induction agent for cesarean section and also to provide analgesia during labor in intermittent boluses.

ELIGIBILITY:
Inclusion criteria:

The study will include 80 ASA physical status I, II patients with age between 18- 50 years old scheduled for elective myomectomy under general anesthesia

Exclusion criteria:

Patients who refused to participate, ASA physical status III, IV, patients younger than 18 years or > 50 years old, BMI > 30, history of epilepsy. Patients having a history of parenteral or oral analgesics within the last 24 hours before initiation of operation or those having allergy to study agents will be excluded.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — opration un female only
Enrollment: 80 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
total Amount of Morphine need intraoperative and postoperative | up to 24 hours
  adjusted to keep the HR and mean arterial blood pressure within 20% of the pre induction values. Starting from the induction till the end of the operation.

SECONDARY OUTCOMES:
duration of surgery | UP TO 1 HOURE
  time from start to end
postoperative pain score | up to 24 hours
  assessment of patient by VAS sore 0= no pain , 10= sever pain
Number of Participants with hallucinations | up to 24 hours
  complication
Number of Participants with sleep disturbances | up to 24 hours
  complication
Number of Participants with nausea and vomiting | up to 24 hour
  complication
Number of Participants with sedation | up to 24 hour
  complication

CONTACTS AND LOCATIONS:
Overall Officials: amr wahadan, MD, Principal Investigator — lecture
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working